CLINICAL TRIAL: NCT06132217
Title: A Phase I/II Study To Evaluate The Safety, Tolerability, Pharmacokinetic Profile And Preliminary Efficacy Of Simmitinib Plus SG001 in Patients With Advanced Solid Tumors
Brief Title: A Study of Simmitinib Plus SG001 in Advanced Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Runshi Pharmaceutical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HA1818-003
Record Dates: First submitted 2023-11-09; First posted 2023-11-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Dose Escalation Phase Cohort 1 (Experimental)
  Interventions: Drug: Simmitinib; Drug: SG001
- Dose Escalation Phase Cohort 2 (Experimental)
  Interventions: Drug: Simmitinib; Drug: SG001
- Dose Escalation Phase Cohort 3 (Experimental)
  Interventions: Drug: Simmitinib; Drug: SG001
- Dose Expansion Phase Cohort A (Experimental)
  Interventions: Drug: Simmitinib; Drug: SG001
- Dose Expansion Phase Cohort B (Experimental)
  Interventions: Drug: Simmitinib; Drug: SG001
- Dose Expansion Phase Cohort C (Experimental)
  Interventions: Drug: Simmitinib; Drug: SG001

INTERVENTIONS:
Drug: Simmitinib — Patients will oral administration according to study protocol until disease progression, death, unacceptable toxicity, loss of follow-up, withdrawal of consent or other conditions meet the end of treatment criteria.
Drug: SG001 — Patients will receive intravenous infusion of SG001 according to study protocol until disease progression, unacceptable toxicity, meeting the suspension or termination criteria, or up to 24 months in patients without disease progression.

SUMMARY:
This is an open-label Phase I/II trial of simmitinib plus SG001 in patients with advanced solid tumors. Phase I will determine and confirm the maximum tolerated dose (MTD) and recommended phase II dose (RP2D) for simmitinib in combination with SG001 in patients with advanced solid tumors. Phase 2 (Expansion) will evaluate the safety and efficacy of the combination in 3 cohorts at the RP2D from Phase I.

ELIGIBILITY:
Inclusion Criteria:

1. Have fully understood and voluntarily sign the ICF for this study;
2. Age of 18-75 years (inclusive);
3. Dose escalation phase: patients with histologically or cytologically confirmed inoperable or metastatic advanced solid tumors;
4. Dose expansion phase: patients who have failed standard treatment (PD or intolerable toxicity after treatment), have no available standard treatment.According to the previous data, the specific tumor cohort was expanded.
5. In the expansion phase, patients should agree to provide tissue specimens for detection of PD-L1 expression levels and/or MSI or dMMR status;
6. At least one measurable lesion according to RECIST 1.1;
7. Eastern Cooperative Oncology Group (ECOG) performance status (PS) score 0-1;
8. Adequate organ function, defined as:

Neutrophil count (ANC) ≥ 1.5 × 10^9/L; Platelet count (PLT) ≥ 100× 10^9/L; Hemoglobin (Hb) ≥ 90 g/L; Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × upper limit of normal (ULN) (≤ 5.0 × ULN for patients with liver metastases); Serum total bilirubin (TBIL) ≤ 1.5 × ULN; Serum creatinine ≤ 1.5 × ULN; Prothrombin time (PT), activated partial thromboplastin time (APTT), international normalized ratio(INR)≤1.5 × ULN; Thyroid Stimulating Hormone (TSH)≤ULN; Left ventricular ejection fraction (LVEF)≥50%; Male and female patients of childbearing age must agree to take effective contraceptive measures during treatment and within 6 months after the last dose of treatment.

Exclusion Criteria:

1. Patients who have previously received any anti-tumor therapy within 4 weeks prior to the first dose;
2. Urine protein ≥ ++ and 24 h urine protein > 1.0g at screening period;
3. Symptomatic central nervous system (CNS) metastases or meningeal metastases;
4. Patients who have previously received any live attenuated vaccine within 4 weeks before the first use of the study treatment or are expected to received any live attenuated vaccine during the study;
5. History of allergic reactions attributed to any monoclonal antibody, and uncontrolled history of allergic asthma;
6. Patients with other types of malignant tumors within 5 years prior to the screening, except for radically resected, non-recurrent skin basal cell carcinoma, skin squamous cell carcinoma, superficial bladder cancer, cervical cancer in situ, or other carcinoma in situ;
7. Patients with any active autoimmune disease requiring systemic therapy within 2 years prior to the first dose;
8. Patients with bleeding tendency; active bleeding or a history of heavy bleeding within the past 6 months;
9. Presence of any severe and/or uncontrolled disease before starting treatment;
10. Any active infection requiring antibiotics or hormones systemic treatment by intravenous infusion within 14 days prior to the first dose;
11. Dose expansion phase: Prior systemic therapy with immunosuppressants or immunoagonists targeting PD-1, PD-L1, CTLA-4, etc;
12. Dose expansion phase: Prior systemic therapy with Antiangiogenic drugs including Anlotinib, Afatinib , Lenvatinib, Sorafenib and Fruquintinib, etc;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2024-01-30 (Estimated); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation Phase: Dose Limited Toxicity (DLT) | From Cycle 1 Day 1 to Cycle 1 Day 28(each cycle is 28 days)
Dose Escalation Phase: Maximum Tolerated Dose (MTD) | From Cycle 1 Day 1 to Cycle 1 Day 28(each cycle is 28 days)
Dose Escalation Phase: Recommended Phase 2 Dose (RP2D) | From Cycle 1 Day 1 to Cycle 1 Day 28(each cycle is 28 days)
Dose Escalation Phase-Incidence rate of Adverse Event (AE). | From first dose to 30 days post the last dose, with approximately 3 years
Dose Expansion Phase - Objective Response Rate (ORR) evaluated by Independent Review Committee (IRC) or investigators in advanced solid tumor based on RECIST 1.1. | Up to approximately 3 years.

SECONDARY OUTCOMES:
Plasma Concentration of simmitinib . | Up to approximately 3 years.
Plasma Concentration of SG001 | Up to approximately 3 years.
Immunogenicity Assessments for Anti-drug Antibody | Up to approximately 3 years.
Dose Escalation Phase: ORR | Up to approximately 3 years.
Disease Control Rate (DCR) | Up to approximately 3 years.
Progression-free Survival (PFS) | Up to approximately 3 years.
Overall Survival (OS) | Up to approximately 3 years.
Duration of Objective Response (DOR) | Up to Approximately 3 years.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital,Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China